CLINICAL TRIAL: NCT01226771
Title: Ribavirin Loading Dose or Priming and Concentration Targeting for HCV Genotype 1
Acronym: RibaC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eu-nr 2010-018332-41; 2010-018332-41 (EudraCT Number)
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis C
Keywords: hepatitis V virus; genotype 1; ribavirin; interferon; Alternative ribavirin dosing
MeSH Terms: conditions — Hepatitis C | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A ("Loading") (Experimental): PEG-IFN α-2a 180 μg/week plus loading (≥26 mg/kg/day for 2 weeks followed by ≥13 mg/kg/day) and concentration targeted (≥ 2.5 mg/L, i.e ≥ 10.25 μmol/L, as measured after 4 weeks of therapy) dosing of ribavirin and response guided treatment duration (RVR 24 weeks, non-RVR 48 weeks, pEVR consider 72 weeks), follow-up period 24 weeks
  Interventions: Drug: Ribavirin "loading" dose given
- Group B ("Priming") (Experimental): Standard-of-care dosing of ribavirin (≥13 mg/kg/day) without PEG-IFN for 4 weeks followed by 24-48 additional weeks of PEG-IFN α-2a 180 μg/week plus standard-of-care dosing of ribavirin (≥13 mg/kg/day) and concentration targeted (≥ 2.5 mg/L, i.e ≥ 10.25 μmol/L, as measured after 28 days after the initiation of ribavirin) dosing of ribavirin and response guided treatment duration (RVR 28 weeks, non-RVR 52 weeks, pEVR consider 76 weeks), follow-up period 24 weeks
  Interventions: Drug: "Priming" dose of ribavirin given
- Group C ("Standard-of-Care) (Active Comparator): PEG-IFN α-2a 180 μg/week plus standard-of-care dosing of ribavirin (≥13 mg/kg/day without any measurement of ribavirin concentration) and response guided treatment duration (RVR 24 weeks, non-RVR 48 weeks, pEVR consider 72 weeks), follow-up period 24 weeks
  Interventions: Drug: Group C ("Standard-of-Care")

INTERVENTIONS:
Drug: Ribavirin "loading" dose given — PEG-IFN α-2a 180 μg/week plus loading (≥26 mg/kg/day for 2 weeks followed by ≥13 mg/kg/day) and concentration targeted (≥ 2.5 mg/L, i.e ≥ 10.25 μmol/L, as measured after 4 weeks of therapy) dosing of ribavirin and response guided treatment duration (RVR 24 weeks, non-RVR 48 weeks, pEVR consider 72 weeks), follow-up period 24 weeks
  Arms: Group A ("Loading")
Drug: "Priming" dose of ribavirin given — Standard-of-care dosing of ribavirin (≥13 mg/kg/day) without PEG-IFN for 4 weeks followed by 24-48 additional weeks of PEG-IFN α-2a 180 μg/week plus standard-of-care dosing of ribavirin (≥13 mg/kg/day) and concentration targeted (≥ 2.5 mg/L, i.e ≥ 10.25 μmol/L, as measured after 28 days after the initiation of ribavirin) dosing of ribavirin and response guided treatment duration (RVR 28 weeks, non-RVR 52 weeks, pEVR consider 76 weeks), follow-up period 24 weeks
  Arms: Group B ("Priming")
Drug: Group C ("Standard-of-Care") — PEG-IFN α-2a 180 μg/week plus standard-of-care dosing of ribavirin (≥13 mg/kg/day without any measurement of ribavirin concentration) and response guided treatment duration (RVR 24 weeks, non-RVR 48 weeks, pEVR consider 72 weeks), follow-up period 24 weeks
  Arms: Group C ("Standard-of-Care)

SUMMARY:
This is a randomized, open-label, parallel group, multicenter pilot study evaluating the efficacy and safety of alternative dosing of ribavirin vs. standard of care dosing in combination with peginterferon alpha-2a in interferon naïve patients with chronic hepatitis c genotype 1 infection.

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate the efficacy and safety of (A) 2 weeks of high dose of ribavirin ("loading", ≥26 mg/kg/day for 14 days followed by ≥13 mg/kg/day) followed by concentration targeted (≥ 2.5 mg/L (10.25 μmol/L) 28 days after initiation of ribavirin therapy) dosing of ribavirin vs. (B) 4 weeks of ribavirin dosing before initiation of PEG-interferon dosing ("priming", ≥13 mg/kg/day) followed by concentration targeted (≥ 2.5 mg/L (10.25 μmol/L) 28 days after initiation of ribavirin therapy) dosing of ribavirin in combination with peginterferon alpha-2a in interferon naïve patients with chronic hepatitis C (CHC) virus genotype 1 infection as compared to (C) standard-of-care dosing of ribavirin (≥13 mg/kg/day without monitoring of ribavirin concentrations) in combination with peginterferon alpha-2a.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients ≥18 years of age
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Serum HCV-RNA ≥15 IU/mL.
* HCV genotype 1 infection confirmed within the past 2 years preceding the initiation of test drug dosing.
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Patients with cirrhosis or transition to cirrhosis must have an abdominal ultrasound, CT scan, or MRI scan without evidence of hepatocellular carcinoma and a serum AFP ≤100 ng/mL within 2 months of randomization
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using effective contraception during treatment and during 4 months for female patients / 7 months for male patients after end of treatment
* Subject must weigh between 45 and 105 kg at screening

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* IFN/ peg-interferon with or without ribavirin therapy at any previous time
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) *6 months prior to the first dose of study drug
* Any investigational drug ≤6 weeks prior to the first dose of study drug.
* HCV genotype 2, 3, 4, 5, 6, or 7 infection.
* Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, anti-HIV Ab
* Evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History or other evidence of decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Serum creatinine level >2 mg/dl (>124 µmol/L) or creatinine clearance ≤50 ml/minute at screening
* Severe psychiatric disease, especially depression, as judged by the treating physician.
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, severe chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Thyroid dysfunction not adequately controlled (TSH and T4 levels out of normal range)
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration) or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension
* Evidence of drug abuse (including excessive alcohol consumption) in accordance with local therapeutic traditions.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Ηemoglobin <12 g/dL in women or <13 g/dL in men at screening.
* Any patient with an increased baseline risk for anemia (e.g. thalassemia major, spherocytosis, history of GI bleeding, etc) or for whom anemia would be medically problematic coagulopathia.
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated
* Evidence of allergy to PEG-IFN or ribavirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The early virological response as measured by decline in HCV-RNA during the first 12 weeks of peginterferon alpha-2a and ribavirin therapy in the three study arms. | The first 12 weeks of therapy

SECONDARY OUTCOMES:
VRVR, RVR, cEVR, pEVR, SVR, and Relapse rates | Throughout the treatment period including 24 weeks post completion of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Infectious Diseases, Gothenburg, Sweden

REFERENCES:
- [Derived] Waldenstrom J, Westin J, Nystrom K, Christensen P, Dalgard O, Farkkila M, Lindahl K, Nilsson S, Norkrans G, Krarup H, Norrgren H, Rauning Buhl M, Stenmark S, Lagging M. Randomized Trial Evaluating the Impact of Ribavirin Mono-Therapy and Double Dosing on Viral Kinetics, Ribavirin Pharmacokinetics and Anemia in Hepatitis C Virus Genotype 1 Infection. PLoS One. 2016 May 11;11(5):e0155142. doi: 10.1371/journal.pone.0155142. eCollection 2016. PMID 27167219